CLINICAL TRIAL: NCT00081705
Title: Estrogen Receptor Variants, HDL, and Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1249; R01HL072941 (NIH)
Record Dates: First submitted 2004-04-19; First posted 2004-04-21 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Arteriosclerosis; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Artery Disease; Heart Diseases

SUMMARY:
To measure the association between estrogen receptor variants and the extent of atherosclerosis in the thoracic and abdominal aorta and the right coronary artery in subjects in the PDAY study.

DETAILED DESCRIPTION:
BACKGROUND:

Increased levels of HDL cholesterol are associated with lower rates of clinical and anatomic atherosclerosis, even in adolescents and young adults. In premenopausal women, estrogen-associated increases in HDL may account for their low rates of coronary heart disease (CHD) events. Recently, a sequence variant in the estrogen receptor-alpha (ER-alpha) gene, ER-alpha IVS1-397 T/C), has been linked to twofold greater increases in HDL cholesterol in response to hormone replacement therapy (HRT). However, it remains unclear whether this sequence variant also augments HDL levels in the setting of premenopausal estrogen exposure and whether such differences translate into greater reductions in atherosclerosis risk. The study uses the cohort of the Pathobiology of Atherosclerosis in Youth (PDAY) study, a large cross-sectional autopsy study of the extent of atherosclerosis in subjects aged 15 to 34 years. The detailed descriptions of atherosclerotic lesions, combined with data on cardiovascular risk factors and access to tissue for DNA extraction, makes this an ideal cohort in which to examine the association between ER-alpha IVS1-397 genotypes, HDL levels, and development of early atherosclerosis.

DESIGN NARRATIVE:

The overall goal for this study is to measure the association between the estrogen receptor (ER- IVS1-401 T/C) polymorphism and extent of abdominal aorta, thoracic artery, and right coronary artery atherosclerosis in Pathobiological Determinants of Atherosclerosis in Youth (PDAY) subjects. The investigators will use DNA extracted from liver specimens in order to measure the ER polymorphisms. The extent of atherosclerosis will be defined as the percent of intimal area involved with fatty streaks or raised lesions, using previously established PDAY definitions. However, percent involvement of fatty streaks alone and the percent involvement of the individual components of raised lesions (fibrous plaques, complicated lesions, and calcified lesions) will be analyzed separately. Available data on risk factors (smoking, diabetes, hyperlipidemia, hypertension) will permit reducing confounding of the results by allowing adjustments for effects of the major risk factors for coronary heart disease. The Department of Pathology at Louisiana State University Health Sciences Center (LSUHSC) has been designated by the National Heart, Lung and Blood Institute to centralize, maintain, and distribute the valuable material collected through the combined efforts of the cooperating institutions for further studies in atherosclerosis. LSUHSC will provide DNA for polymorphism analysis and assist in data analysis. Polymorphism determination will occur at Wake Forest.

ELIGIBILITY:
No eligibility criteria

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Herrington — Wake Forest University Health Sciences